CLINICAL TRIAL: NCT00623467
Title: A Multicenter, Open-label, Phase 3 Study to Determine the Safety and Efficacy of Gadobutrol 1.0 Molar (Gadavist) in Patients Referred for Contrast-enhanced MRI of the Central Nervous System (CNS).
Brief Title: Safety and Efficacy of Gadobutrol 1.0 Molar ( Gadavist ) in Patients for Central Nervous System (CNS) Imaging
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 91682
Record Dates: First submitted 2008-02-18; First posted 2008-02-26 (Estimated); Results first posted 2011-10-06 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-01

CONDITIONS: Central Nervous System Diseases
Keywords: Central Nervous System Imaging; Diagnostic Imaging
MeSH Terms: conditions — Central Nervous System Diseases | interventions — gadobutrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gadobutrol (Gadavist, BAY86-4875) (Experimental): Participants were administered a single dose of gadobutrol 0.1 mmol/kg body weight (bw) via i.v. (intravenous) bolus administration using a power injector via a peripheral vein (an antecubital vein was preferred). Gadobutrol was injected at a rate of 2 mL/second followed by a 20-mL 0.9% saline flush at the same rate.
  Interventions: Drug: Gadobutrol (Gadavist, Gadovist, BAY86-4875)

INTERVENTIONS:
Drug: Gadobutrol (Gadavist, Gadovist, BAY86-4875) — Gadobutrol single injection 0.1 mmol/kg BW via IV bolus administration at 2mL/sec.

SUMMARY:
This is a study involving the use of Magnetic Resonance Imaging (MRI) contrast agents called Gadavist. The purpose of this study is to look at the safety (what are the side effects) and efficacy (how well does it work) of Gadavist when used for taking images of the brain and spine. The results of the MRI will be compared to the results of images taken without Gadavist.

DETAILED DESCRIPTION:
Issues on safety will be addressed in Adverse Events section.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for contrast enhanced MRI of the CNS based on symptoms or previous procedures.

Exclusion Criteria:

* Patients with acute renal insufficiency
* Patients with severe renal disease
* Patients with any contraindication to magnetic resonance imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2007-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (37):
- United States (21):
  - HOPE Research Institute, LLC, Phoenix, Arizona
  - Scottsdale Medical Imaging, Ltd., Scottsdale, Arizona
  - Radiology Ltd., Tucson, Arizona
  - Landmark Imaging Medical Group, Los Angeles, California
  - Cedars- Sinai Medical Center, Los Angeles, California
  - Sharp & Children's MRI Center, San Diego, California
  - University of Florida - Jacksonville, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - River Birch Research Alliance, LLC, Blue Ridge, Georgia
  - Eisenhower Army Medical Center, Fort Gordon, Georgia
  - University of Michigan Health System, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Bio-Magnetic Resonance, Inc., Madison Heights, Michigan
  - Maimonides Medical Center, Brooklyn, New York
  - Mount Sinai Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor College of Medicine, Houston, Texas
- Argentina (4):
  - Investigaciones Médicas, Buenos Aires, Ciudad Auton. de Buenos Aires
  - Milbet Diagnostico por Imagenes, Buenos Aires, Ciudad Auton. de Buenos Aires
  - Hospital Italiano Buenos Aires, Buenos Aires, Ciudad Auton. de Buenos Aires
  - Centro de Diagnóstico Dr. Enrique Rossi, Buenos Aires, Ciudad Auton. de Buenos Aires
- China (5):
  - Zhongda Hosp. affiliated of Southeast Univ., Nanjing, Jiangsu
  - The 1st Affiliated Hosp of the 4th Military Med Uni, Xi'an, Shaanxi
  - Chinese PLA General Hosp., Beijing
  - Affiliated Ruijin Hosp. Shanghai Jiaotong Univ. Med School, Shanghai
  - Fudan University Huashan Hospital, Shanghai
- Colombia (2):
  - Fundación Instituto de Alta tecnología médica de Antioquia, Medellín, Antioquia
  - Fundación Santa Fe de Bogotá - Hospital Universitario, Bogotá, Cundinamarca
- South Korea (5):
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul, Korea
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University College of Medicine, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The date of the first participant's first visit was 17 DEC 2007. The date of the last participant's last visit was 12 DEC 2008.
Pre-assignment Details: A total of 347 participants were screened for inclusion into the study; 4 participants failed screening because they did not meet the inclusion criteria. Therefore, 343 participants were enrolled into the study and received study drug.
Period: Overall Study
Arm/Group | Gadobutrol (Gadavist, BAY86-4875)
Started | 343
Completed | 336
Not Completed | 7
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 4
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 343
Age, Customized [Number; unit: participants]
  < 45 years | 149
  45 - 64 years | 145
  ≥ 65 years | 49
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197
  Male | 146
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 68
  Black | 9
  Hispanic | 87
  Asian | 161
  Other | 18

OUTCOME MEASURES:

1. Primary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Combined Unenhanced/Gadobutrol-enhanced Magnetic Resonance Imaging (MRI) Compared to Unenhanced MRI by Blinded Reader 1 (BR1)
Description: BR1 (reader 1 of 3) evaluated the images from the unenhanced magnetic resonance imaging (MRI) in one session and the images from the combined unenhanced and gadobutrol-enhanced MRIs in another. Contrast enhancement was scored on a 4-point scale where 1 = no enhancement and 4 = excellent enhancement. Border delineation was scored on a 4-point scale where 1 = no or unclear delineation and 4 = excellent delineation. Internal morphology was scored on a 3-point scale where 1 = poorly visible and 3 = sufficiently visible.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: The full analysis set (FAS); which used data from all participants for whom data and images were available for the unenhanced MRI and combined unenhanced and gadobutrol-enhanced MRI, excluding the sample participants (the first participant from each study site).
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Unenhanced: Participants had diagnostic imaging before receiving any contrast agent
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 301 | 301
scores on a scale
  contrast enhancement | 0.94 (0.25) | 2.96 (0.80)
  border delineation | 2.17 (0.57) | 3.01 (0.75)
  internal morphology | 1.87 (0.51) | 2.40 (0.54)
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t-test — for contrast enhancement; Mean Difference (Final Values) = 2.03, Standard Deviation 0.86
Statistical Analysis 2: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Final Values) = 0.85, Standard Deviation 0.74
Statistical Analysis 3: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.53, Standard Deviation 0.54

2. Primary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Combined Unenhanced/Gadobutrol-enhanced Magnetic Resonance Imaging (MRI) Compared to Unenhanced MRI by Blinded Reader 2 (BR2)
Description: BR2 (reader 2 of 3) evaluated the images from the unenhanced MRI in one session and the images from the combined unenhanced and gadobutrol-enhanced MRIs in another. Contrast enhancement was scored on a 4-point scale where 1 = no enhancement and 4 = excellent enhancement. Border delineation was scored on a 4-point scale where 1 = no or unclear delineation and 4 = excellent delineation. Internal morphology was scored on a 3-point scale where 1 = poorly visible and 3 = sufficiently visible.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 309 | 309
scores on a scale
  contrast enhancement | 0.93 (0.27) | 2.87 (0.77)
  border delineation | 1.98 (0.56) | 3.15 (0.73)
  internal morphology | 1.38 (0.43) | 2.46 (0.54)
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t-test — for contrast enhancement; Mean Difference (Final Values) = 1.94, Standard Deviation 0.80
Statistical Analysis 2: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Final Values) = 1.17, Standard Deviation 0.94
Statistical Analysis 3: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 1.08, Standard Deviation 0.74

3. Primary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Combined Unenhanced/Gadobutrol-enhanced Magnetic Resonance Imaging (MRI) Compared to Unenhanced MRI by Blinded Reader 3 (BR3)
Description: BR3 (reader 3 of 3) evaluated the images from the unenhanced MRI in one session and the images from the combined unenhanced and gadobutrol-enhanced MRIs in another. Contrast enhancement was scored on a 4-point scale where 1 = no enhancement and 4 = excellent enhancement. Border delineation was scored on a 4-point scale where 1 = no or unclear delineation and 4 = excellent delineation. Internal morphology was scored on a 3-point scale where 1 = poorly visible and 3 = sufficiently visible.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 309 | 309
scores on a scale
  contrast enhancement | 0.93 (0.25) | 2.86 (0.77)
  border delineation | 1.64 (0.45) | 2.76 (0.76)
  internal morphology | 1.49 (0.39) | 2.25 (0.56)
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t-test — for contrast enhancement; Mean Difference (Final Values) = 1.93, Standard Deviation 0.82
Statistical Analysis 2: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Net) = 1.12, Standard Deviation 0.74
Statistical Analysis 3: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.77, Standard Deviation 0.57

4. Primary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Combined Unenhanced/Gadobutrol-enhanced Magnetic Resonance Imaging (MRI) Compared to Unenhanced MRI by Average Reader (AR)
Description: The AR analysis used the mean of the values for the 3 blinded readers. The 3 BRs evaluated the images from the unenhanced MRI in one session and the images from the combined unenhanced and gadobutrol-enhanced MRIs in another. Contrast enhancement was scored on a 4-point scale where 1 = no enhancement and 4 = excellent enhancement. Border delineation was scored on a 4-point scale where 1 = no or unclear delineation and 4 = excellent delineation. Internal morphology was scored on a 3-point scale where 1 = poorly visible and 3 = sufficiently visible.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 311 | 311
scores on a scale
  contrast enhancement | 0.93 (0.23) | 2.86 (0.73)
  border delineation | 1.92 (0.43) | 2.94 (0.68)
  internal morphology | 1.57 (0.35) | 2.35 (0.49)
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t-test — for contrast enhancement; Mean Difference (Final Values) = 1.94, Standard Deviation 0.77
Statistical Analysis 2: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Final Values) = 1.02, Standard Deviation 0.71
Statistical Analysis 3: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.78, Standard Deviation 0.53

5. Primary Outcome: Number of Lesions for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Blinded Readers
Description: The 3 blinded readers evaluated the images from the unenhanced MRI in one session and the images from the combined unenhanced and gadobutrol-enhanced MRIs in another to determine the total number of lesions.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: FAS
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 321 | 321
lesions
  BR1 | 2.26 (7.61) | 2.93 (8.68)
  BR2 | 3.77 (11.79) | 3.60 (10.40)
  BR3 | 1.92 (7.19) | 2.37 (7.26)
  AR | 2.65 (6.30) | 2.97 (6.95)
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; Mean Difference (Final Values) = 0.66, Standard Deviation 5.31 — for BR1
Statistical Analysis 2: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; Mean Difference (Final Values) = -0.17, Standard Deviation 8.77 — for BR2
Statistical Analysis 3: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; Mean Difference (Final Values) = 0.45, Standard Deviation 4.20 — for BR3
Statistical Analysis 4: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Non-Inferiority or Equivalence — noninferiority margin = -0.35; 95% confidence interval for paired means; Mean Difference (Final Values) = 0.32, 95% CI 2-sided [-0.070 to 0.704], Standard Deviation 3.53 — confidence interval provided for average reader, lower limit is compared to noninferiority margin

6. Secondary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Clinical Investigator
Description: The clinical investigators evaluated the images from the unenhanced MRI in one session and the images from the combined unenhanced and gadobutrol-enhanced MRIs in another. Contrast enhancement was scored on a 4-point scale where 1 = no enhancement and 4 = excellent enhancement. Border delineation was scored on a 4-point scale where 1 = no or unclear delineation and 4 = excellent delineation. Internal morphology was scored on a 3-point scale where 1 = poorly visible and 3 = sufficiently visible. The data for "contrast enhancement - unenhanced" were not collected for the clinical investigators.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 312 | 312
scores on a scale
  contrast enhancement | NA (NA) — The data for "contrast enhancement - unenhanced" were not collected for the clinical investigators. | 2.97 (0.80)
  border delineation | 2.51 (0.75) | 3.40 (0.50)
  internal morphology | 2.03 (0.64) | 2.78 (0.30)
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t-test — for border delineation; Mean Difference (Final Values) = 0.89, Standard Deviation 0.68
Statistical Analysis 2: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.74, Standard Deviation 0.65

7. Secondary Outcome: Number of Lesions for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Clinical Investigator
Description: The clinical investigators evaluated the images from the unenhanced MRI in one session and the images from the combined unenhanced and gadobutrol-enhanced MRIs in another to determine the total number of lesions.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: FAS
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 321 | 321
lesions | 2.53 (4.60) | 2.74 (4.78)
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Non-Inferiority or Equivalence — noninferiority margin = -0.35; Mean Difference (Final Values) = 0.21, 95% CI [0.030 to 0.381], Standard Deviation 1.60 — lower limit of the confidence interval is compared to the noninferiority margin

8. Secondary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Lesions for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Blinded Reader 1 (BR1)
Description: BR1 (reader 1 of 3) evaluated the images from the unenhanced MRI in one session and the images from the combined unenhanced and gadobutrol-enhanced MRIs in another. Contrast enhancement was scored on a 4-point scale where 1 = no enhancement and 4 = excellent enhancement. Border delineation was scored on a 4-point scale where 1 = no or unclear delineation and 4 = excellent delineation. Internal morphology was scored on a 3-point scale where 1 = poorly visible and 3 = sufficiently visible.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 245 | 245
scores on a scale
  contrast enhancement | 0.84 (0.40) | 2.42 (1.37)
  border delineation | 1.66 (0.96) | 2.40 (1.15)
  internal morphology | 1.66 (0.94) | 2.11 (0.88)
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t-test — for contrast enhancement; Mean Difference (Final Values) = 1.59, Standard Deviation 1.47
Statistical Analysis 2: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Final Values) = 0.75, Standard Deviation 1.34
Statistical Analysis 3: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.45, Standard Deviation 1.03

9. Secondary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Lesions for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Blinded Reader 2 (BR2)
Description: as for outcome 2
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 246 | 246
scores on a scale
  contrast enhancement | 0.80 (0.42) | 2.28 (1.26)
  border delineation | 1.67 (0.98) | 2.79 (1.21)
  internal morphology | 1.19 (0.74) | 2.22 (0.91)
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t-test — for contrast enhancement; Mean Difference (Final Values) = 1.49, Standard Deviation 1.38
Statistical Analysis 2: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Final Values) = 1.12, Standard Deviation 1.60
Statistical Analysis 3: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 1.02, Standard Deviation 1.25

10. Secondary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Lesions for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Blinded Reader 3 (BR3)
Description: as for outcome 3
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 248 | 248
scores on a scale
  contrast enhancement | 0.81 (0.41) | 2.48 (1.29)
  border delineation | 1.07 (0.71) | 2.34 (1.22)
  internal morphology | 1.10 (0.70) | 2.00 (0.93)
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t-test — for contrast enhancement; Mean Difference (Final Values) = 1.67, Standard Deviation 1.39
Statistical Analysis 2: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Final Values) = 1.26, Standard Deviation 1.30
Statistical Analysis 3: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.91, Standard Deviation 1.02

11. Secondary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Lesions for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Average Reader (AR)
Description: as for outcome 4
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 273 | 273
scores on a scale
  contrast enhancement | 0.79 (0.38) | 2.29 (1.23)
  border delineation | 1.42 (0.77) | 2.42 (1.08)
  internal morphology | 1.27 (0.68) | 2.04 (0.82)
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t-test — for contrast enhancement; Mean Difference (Final Values) = 1.51, Standard Deviation 1.32
Statistical Analysis 2: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Final Values) = 1.00, Standard Deviation 1.27
Statistical Analysis 3: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.77, Standard Deviation 0.99

12. Secondary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Normal Structures for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Blinded Reader 1 (BR1)
Description: as for outcome 8
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 289 | 289
scores on a scale
  contrast enhancement | 1.00 (0.04) | 3.40 (0.48)
  border delineation | 2.57 (0.45) | 3.51 (0.49)
  internal morphology | 2.03 (0.30) | 2.65 (0.35)
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t-test — for contrast enhancement; Mean Difference (Final Values) = 2.40, Standard Deviation 0.48
Statistical Analysis 2: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Final Values) = 0.93, Standard Deviation 0.46
Statistical Analysis 3: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.62, Standard Deviation 0.32

13. Secondary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Normal Structures for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Blinded Reader 2 (BR2)
Description: as for outcome 2
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 289 | 289
scores on a scale
  contrast enhancement | 1.01 (0.09) | 3.36 (0.39)
  border delineation | 2.18 (0.29) | 3.45 (0.38)
  internal morphology | 1.49 (0.22) | 2.67 (0.27)
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t-test — for contrast enhancement; Mean Difference (Final Values) = 2.35, Standard Deviation 0.40
Statistical Analysis 2: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Final Values) = 1.27, Standard Deviation 0.38
Statistical Analysis 3: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 1.17, Standard Deviation 0.34

14. Secondary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Normal Structures for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Blinded Reader 3 (BR3)
Description: as for outcome 3
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 289 | 289
scores on a scale
  contrast enhancement | 1.00 (0.05) | 3.22 (0.37)
  border delineation | 2.07 (0.27) | 3.15 (0.38)
  internal morphology | 1.79 (0.16) | 2.50 (0.27)
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t-test — for contrast enhancement; Mean Difference (Final Values) = 2.21, Standard Deviation 0.37
Statistical Analysis 2: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Final Values) = 1.07, Standard Deviation 0.45
Statistical Analysis 3: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.72, Standard Deviation 0.30

15. Secondary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Normal Structures for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Average Reader (AR)
Description: as for outcome 4
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 289 | 289
scores on a scale
  contrast enhancement | 1.01 (0.04) | 3.33 (0.34)
  border delineation | 2.28 (0.27) | 3.37 (0.34)
  internal morphology | 1.77 (0.15) | 2.61 (0.24)
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t-test — for contrast enhancement; Mean Difference (Final Values) = 2.32, Standard Deviation 0.34
Statistical Analysis 2: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t test — for border delineation; Mean Difference (Final Values) = 1.09, Standard Deviation 0.30
Statistical Analysis 3: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.84, Standard Deviation 0.22

16. Secondary Outcome: Scores for Contrast Enhancement for Lesions for Combined Unenhanced/Gadobutrol-enhanced MRI by Clinical Investigator
Description: The clinical investigators evaluated the images from the combined unenhanced and gadobutrol-enhanced MRIs. Contrast enhancement was scored on a 4-point scale where 1 = no enhancement and 4 = excellent enhancement. The data for contrast enhancement - gadobutrol combined was shown below.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 284
scores on a scale | 2.84 (1.24)

17. Secondary Outcome: Scores for Two Visualization Parameters (Border Delineation and Internal Morphology) for Lesions for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Clinical Investigator
Description: The clinical investigators evaluated the images from the unenhanced MRI in one session and the images from the combined unenhanced and gadobutrol-enhanced MRIs in another. Border delineation was scored on a 4-point scale where 1 = no or unclear delineation and 4 = excellent delineation. Internal morphology was scored on a 3-point scale where 1 = poorly visible and 3 = sufficiently visible.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 285 | 285
scores on a scale
  border delineation | 2.44 (1.01) | 3.26 (0.79)
  internal morphology | 2.06 (0.82) | 2.73 (0.50)
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t-test — for border delineation; Mean Difference (Final Values) = 0.82, Standard Deviation 1.00
Statistical Analysis 2: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.66, Standard Deviation 0.90

18. Secondary Outcome: Scores for Three Visualization Parameters (Contrast Enhancement, Border Delineation and Internal Morphology) for Normal Structures for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Clinical Investigator
Description: The clinical investigators evaluated the images from the unenhanced MRI in one session and the images from the combined unenhanced and gadobutrol-enhanced MRIs in another. Contrast enhancement was scored on a 4-point scale where 1 = no enhancement and 4 = excellent enhancement. Border delineation was scored on a 4-point scale where 1 = no or unclear delineation and 4 = excellent delineation. Internal morphology was scored on a 3-point scale where 1 = poorly visible and 3 = sufficiently visible.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 289 | 289
scores on a scale
  contrast enhancement | NA (NA) — The data for "contrast enhancement - unenhanced" were not collected for the clinical investigators. | 3.47 (0.50)
  border delineation | 2.56 (0.69) | 3.55 (0.41)
  internal morphology | 1.97 (0.65) | 2.82 (0.25)
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t-test — for border delineation; Mean Difference (Final Values) = 0.99, Standard Deviation 0.63
Statistical Analysis 2: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t test — for internal morphology; Mean Difference (Final Values) = 0.85, Standard Deviation 0.64

19. Secondary Outcome: Percentage (Per.) of the Exact Diagnostic Matches (Accuracy of Diagnosis) for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Majority Reader
Description: The majority reader diagnosis was the diagnosis provided by at least 2 of the BRs. The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. The accuracy of the majority reader diagnoses for the combined unenhanced/gadobutrol-enhanced and the unenhanced MR images was the percentage of the exact matches with the final clinical diagnosis.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: per. of the exact diagnostic matches
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 224 | 224
per. of the exact diagnostic matches | 51.8 | 61.2
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p = 0.0002, McNemar; Risk Difference (RD) = 9.4

20. Secondary Outcome: Percentage (Per.) of the Exact Diagnostic Matches (Accuracy of Diagnosis) for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Clinical Investigator
Description: The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. The accuracy of the investigator diagnoses for the combined unenhanced/gadobutrol-enhanced and the unenhanced MR images was the percentage of the exact matches with the final clinical diagnosis.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: per. of the exact diagnostic matches
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 261 | 261
per. of the exact diagnostic matches | 67.0 | 74.3
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p = 0.0001, McNemar; Risk Difference (RD) = 7.3

21. Secondary Outcome: Accuracy of Detection of Normal/Abnormal Brain Tissue for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Majority Reader Using T1-weighted (T1w) Images
Description: The majority reader diagnosis was the diagnosis provided by at least 2 of the 3 BRs for the T1w assessment (normal or abnormal). The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. Accuracy = percentage of participants for which the imaging modality (unenhanced or Gadobutrol-enhanced) matches the standard of truth for the presence or absence of abnormal brain tissue.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 239 | 239
percentage of participants | 74.9 | 79.9
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p = 0.0285, McNemar; Risk Difference (RD) = 5.0

22. Secondary Outcome: Sensitivity of Detection of Normal/Abnormal Brain Tissue for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Majority Reader Using T1-weighted (T1w) Images
Description: The majority reader diagnosis was the diagnosis provided by at least 2 of the 3 BRs for the T1w assessment (normal or abnormal). The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. Sensitivity = percentage of participants for which the imaging modality (unenhanced or Gadobutrol-enhanced) correctly detects abnormal brain tissue as defined by the independent truth committee.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 199 | 199
percentage of participants | 75.4 | 83.9
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p = 0.0004, McNemar; Risk Difference (RD) = 8.5

23. Secondary Outcome: Specificity of Detection of Normal/Abnormal Brain Tissue for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Majority Reader Using T1-weighted (T1w) Images
Description: The majority reader diagnosis was the diagnosis provided by at least 2 of the 3 BRs for the T1w assessment (normal or abnormal). The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. Specificity = percentage of participants for which the imaging modality (unenhanced or Gadobutrol-enhanced) correctly excludes abnormal brain tissue as defined by the independent truth committee
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 40 | 40
percentage of participants | 72.5 | 60.0
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p = 0.0588, McNemar; Risk Difference (RD) = -12.5

24. Secondary Outcome: Accuracy of Detection of Malignant Lesions (ML) for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Majority Reader
Description: The presence of malignant lesions was derived from the diagnoses given on the evaluation of the unenhanced image set and the combined unenhanced/enhanced image sets. The majority reader diagnosis was the diagnosis provided by at least 2 of the 3 BRs. The final clinical diagnosis was provided by an independent truth committee not using the study-specific MR image sets. Accuracy = percentage of participants for which the imaging modality (unenhanced or Gadobutrol-enhanced) matches the standard of truth for the presence or absence of malignant lesions.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 261 | 261
percentage of participants | 82.4 | 87.4
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p = 0.0093, McNemar; Risk Difference (RD) = 5.0

25. Secondary Outcome: Sensitivity of Detection of Malignant Lesions (ML) for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Majority Reader
Description: The presence of malignant lesions was derived from the diagnoses given on the evaluation of the unenhanced image set and the combined unenhanced/enhanced image sets. The majority reader diagnosis was the diagnosis provided by at least 2 of the 3 BRs. The final clinical diagnosis was provided by an independent truth committee not using the study-specific MR image sets. Sensitivity = percentage of participants for which the imaging modality (unenhanced or Gadobutrol-enhanced) correctly detects malignant lesions as defined by the independent truth committee.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 63 | 63
percentage of participants | 57.1 | 77.8
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p = 0.0003, McNemar; Risk Difference (RD) = 20.6

26. Secondary Outcome: Specificity of Detection of Malignant Lesions (ML) for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Majority Reader
Description: The presence of malignant lesions was derived from the diagnoses given on the evaluation of the unenhanced image set and the combined unenhanced/enhanced image sets. The majority reader diagnosis was the diagnosis provided by at least 2 of the 3 BRs. The final clinical diagnosis was provided by an independent truth committee not using the study-specific MR image sets. Specificity = percentage of participants for which the imaging modality (unenhanced or Gadobutrol-enhanced) correctly excludes malignant lesions as defined by the independent truth committee.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 198 | 198
percentage of participants | 90.4 | 90.4
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p = 1.0000, McNemar; Risk Difference (RD) = 0.0

27. Secondary Outcome: Accuracy of Detection of Malignant Lesions (ML) for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Clinical Investigator
Description: The presence of malignant lesions was derived from the diagnoses given by the investigator on the evaluation of the unenhanced image set and the combined unenhanced/enhanced image sets. The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. Accuracy = percentage of participants for which the imaging modality (unenhanced or Gadobutrol-enhanced) matches the standard of truth for the presence or absence of malignant lesions.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 261 | 261
percentage of participants | 88.9 | 92.7
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p = 0.0016, McNemar; Risk Difference (RD) = 3.8

28. Secondary Outcome: Sensitivity of Detection of Malignant Lesions (ML) for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Clinical Investigator
Description: The presence of malignant lesions was derived from the diagnoses given by the investigator on the evaluation of the unenhanced image set and the combined unenhanced/enhanced image sets. The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. Sensitivity = percentage of participants for which the imaging modality (unenhanced or Gadobutrol-enhanced) correctly detects malignant lesions as defined by the independent truth committee.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 63 | 63
percentage of participants | 71.4 | 79.4
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p = 0.0253, McNemar; Risk Difference (RD) = 7.9

29. Secondary Outcome: Specificity of Detection of Malignant Lesions (ML) for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Clinical Investigator
Description: The presence of malignant lesions was derived from the diagnoses given by the investigator on the evaluation of the unenhanced image set and the combined unenhanced/enhanced image sets. The final clinical diagnosis was provided by an independent truth committee following evaluation of findings from referral through a 3-month follow-up period, not including the study-specific MR image sets. Specificity = percentage of participants for which the imaging modality (unenhanced or Gadobutrol-enhanced) correctly excludes malignant lesions as defined by the independent truth committee.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: All participants in the FAS with assessments for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 198 | 198
percentage of participants | 94.4 | 97.0
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p = 0.0253, McNemar; Risk Difference (RD) = 2.5

30. Secondary Outcome: Diagnostic Confidence for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Average Reader
Description: The BRs recorded his/her confidence in diagnosis for the unenhanced MR image set and the combined unenhanced/enhanced MR image sets. The degree of confidence was rated on a 4-point scale where 1 = not confident and 4 = very confident. The AR score was the mean of the means of the 3 BRs.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 321 | 321
scores on a scale | 2.70 (0.61) | 3.13 (0.64)
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t-test; Mean Difference (Final Values) = 0.44, Standard Deviation 0.70

31. Secondary Outcome: Diagnostic Confidence for Combined Unenhanced/Gadobutrol-enhanced MRI Compared to Unenhanced MRI by Clinical Investigator
Description: The investigator recorded his/her confidence in diagnosis for the unenhanced MR image set and the combined unenhanced/enhanced MR image sets. The degree of confidence was rated on a 4-point scale where 1 = not confident and 4 = very confident.
Time Frame: Up to 2 hours after injection of gadobutrol
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Unenhanced | Gadobutrol (Gadavist, BAY86-4875)
Number analyzed (Participants) | 321 | 321
scores on a scale | 2.61 (0.95) | 3.45 (0.74)
Statistical Analysis 1: Comparison: Unenhanced vs Gadobutrol (Gadavist, BAY86-4875); Test type: Superiority or Other; p < 0.0001, paired t-test; Mean Difference (Final Values) = 0.84, Standard Deviation 0.81

ADVERSE EVENTS:
Arm/Group | Gadobutrol (Gadavist, BAY86-4875)
Serious Adverse Events (participants affected / at risk) | 1/343
Other Adverse Events (participants affected / at risk) | 29/343
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gadobutrol (Gadavist, BAY86-4875) (N=343)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gadobutrol (Gadavist, BAY86-4875) (N=343)
Nausea (Gastrointestinal disorders) | 8 (8)
Fatigue (General disorders) | 5 (5)
Red blood cells urine positive (Investigations) | 4 (4)
White blood cells urine positive (Investigations) | 5 (5)
Headache (Nervous system disorders) | 12 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor is interested in the publication of the results of every study it performs. All relevant aspects regarding publication will be part of the contract between the sponsor and the investigator/institution. The sponsor has committed to the global industry position on disclosure of information about clinical trials. The information regarding the study protocol is made publicly available on the internet at www.clinicaltrials.gov.